CLINICAL TRIAL: NCT01256983
Title: Daily Light Intervention in Renal Transplant Recipients Having a Sleep-Wake Dysregulation
Brief Title: Light for Renal Transplant Recipients Having a Sleep-Wake Dysregulation
Acronym: SleepTx-1
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Zürich (Other)
Responsible Party: Principal Investigator, Hanna Burkhalter, PhD, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SleepTx-1
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Renal Disease; Sleep Disorders
Keywords: Sleep quality; Daytime Sleepiness
MeSH Terms: conditions — Kidney Diseases; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bright Light Therapy (Experimental): Bright Light Therapy with 10000 lux beginning at day 21 until day 42
  Interventions: Behavioral: Bright Light Therapy
- Wait-list intervention (Other): Wait-list design Intervention. Bright Light Therapy with 10000 lux beginning at day 63 until day 84, when the 9 study weeks were over.
  Interventions: Behavioral: Wait-list intervention

INTERVENTIONS:
Behavioral: Bright Light Therapy — 10000 Lux for 30 Minutes according to sleep wake rhythm
  Other Names: Philips Energy Light
  Arms: Bright Light Therapy
Behavioral: Wait-list intervention — 10000 Lux for 30 Minutes according to sleep wake rhythm
  Other Names: Philips Energy Light
  Arms: Wait-list intervention

SUMMARY:
Sleep-wake dysregulation is a disturbance in the roughly 24-hour cycle of the circadian rhythm. Well known disorders presenting a sleep-wake dysregulation are seasonal affective disorder, jet lag and shift work. These people experience a serious mood change when the seasons change. When the day-night rhythm is desynchronized, they have sleep disturbances, little energy, and often feel depressed. An established intervention to treat this disorder is bright light therapy. Light therapy is used for affective disorders for shift workers, jet lag symptomatology and for advancing or delaying desynchronized rhythms.Two proxy measures for sleep-wake dysregulation are sleep quality and daytime sleepiness. It is known from cross sectional studies that renal transplant (RTx) recipients have a prevalence between 30% to 62% of poor sleep quality measured by self report; a prevalence of impaired daytime functioning of 34% 12 and a prevalence of depressive symptomatology of 20% to 22%. Sleep-wake dysregulation in other chronically ill population are a risk factor for morbidity and mortality.

RTx nurses in the follow-up care are in the frontline for recipient's symptoms respectively problems. The psychosocial variables that should be addressed, having an association with morbidity and mortality are sleep, daytime functioning, adherence to immunosuppressive medication, exercise, smoking and depressive symptomatology.

In the following research project we will address the following gaps: the fact that nature of sleep disturbances in RTx recipients has never been assessed, that there is no prevalence available on sleep-wake dysregulation and that there is no data on bright light therapy intervention in RTx recipients.

Hypothesis: Renal transplant recipients having a sleep wake disregulation will have an improved sleep quality and less daytime sleepiness after 21 days of light therapy.

DETAILED DESCRIPTION:
This research project has three phases:

The first phase is a cross sectional survey including all patients transplanted in Basel, Bern and in Zurich speaking German and transplanted at least 6 months ago. Renal transplant recipients having poor sleep quality and / or daytime sleepiness as result of this first phase will be asked to participate in phase two. Phase two is an sleep assessment, resulting in a presumed sleep diagnosis.

Renal transplant recipients having a sleep wake dysregulation, assessed in phase two, will be asked to participate in phase three. Phase three is a pilot randomized controlled trial to compare the sustained impact of bright light therapy on sleep-wake regulation.

ELIGIBILITY:
Inclusion Criteria:

* For phase 1: all renal transplant recipients transplanted at the University Hospital Basel, Bern and Zurich, speaking German and having an actual address on the follow-up list of the ambulatory center list.
* Renal transplant recipients who have poor Sleep quality and /or daytime sleepiness (phase 1: Cross sectional survey study) and had a Sleep assessment (phase 2: Cross sectional diagnostic interview study)
* Renal transplant recipients who participated in Phase 1 and 2 that were diagnosed with sleep wake dysregulation
* Renal transplant recipients with signed written informed consent.

Exclusion Criteria:

* RTx recipients, who participated in phase 2, will be excluded in the study if

  * they were diagnosed with sleep disorders as parasomnia, breathing disorders or movement disorders.
  * they were diagnosed with alcohol or substance abuse
  * they are blind or suffer from a severe vision impairment (cataract), which possibly limits the effect of the light intervention and patients taking photosensitive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabina De De Geest, PhD, Principal Investigator — Institute of Nursing Science

REFERENCES:
- [Derived] Burkhalter H, Wirz-Justice A, Denhaerynck K, Fehr T, Steiger J, Venzin RM, Cajochen C, Weaver TE, De Geest S. The effect of bright light therapy on sleep and circadian rhythms in renal transplant recipients: a pilot randomized, multicentre wait-list controlled trial. Transpl Int. 2015 Jan;28(1):59-70. doi: 10.1111/tri.12443. Epub 2014 Oct 2. PMID 25182079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 patients were recruited
Pre-assignment Details: 19 declined to participate after initial interest
Groups:
- Light Box: 10000 lux after day 21
  Light Box : 10000 Lux for 30 Minutes according to sleep wake rhythm
- No Intervention: 10000 Lux after day 63
Period: Overall Study
Arm/Group | Light Box | No Intervention
Started | 15 | 15
Completed | 14 | 12
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Light Box | No Intervention | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.72 (10.33) | 58.54 (14.91) | 59.63 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  Switzerland | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Bedtime
Description: The mean "bedtime" assessed by actimetry of each 3 week period (day 21, 42, 63 ) was used as outcome to be compared with the control group.
  Bedtime is expressed in time (hours and minutes)
Time Frame: Mean Bedtimes over 21 days for each period
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Light Box | No Intervention
Number analyzed (Participants) | 14 | 12
Hours
  Getup time | 7.44 (1.69) | 7.24 (1.39)
  Bedtime | 22.98 (1.78) | 22.48 (1.37)

ADVERSE EVENTS:
Time Frame: 2 months
Description: 2 months beginning with the start of the study.
Arm/Group | Bright Light Therapy | Wait-list Intervention
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
The study was very long and burdensome for the participants, a full powered study should be shorter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes